CLINICAL TRIAL: NCT03575962
Title: A Single Centre, 2-period, Randomized, Open-label Phase 1 Study to Assess the Relative Bioavailability of a Mesylate Salt Capsule of GSK3640254 Compared to a Hydrochloride Salt Capsule in Healthy Participants
Brief Title: A Study to Compare the Relative Bioavailability of Two Different Formulations of GSK3640254
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 208131; 2018-001175-21 (EudraCT Number)
Record Dates: First submitted 2018-06-12; First posted 2018-07-03 (Actual); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-07

CONDITIONS: HIV Infections
Keywords: 2-period; Pharmacokinetics; FTIH; GSK3640254; healthy subject; bioavailability
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Subjects will receive GSK3640254 bis-hydrochloride salt capsule followed by mesylate salt capsule or vice versa in two treatment periods.
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GSK3640254 Bis-hydrochloride followed by GSK3640254 mesylate (Experimental): The subjects in this arm will receive an oral administration of 200 mg, as 2 GSK3640254 bis-hydrochloride salt Capsules(reference), as single oral dose, on the morning of Day 1 during Period 1 of the study. This will be followed by an oral administration of 200 mg, as 2 GSK3640254 Mesylate salt capsule (test), as single oral dose, on the morning of Day 1, during Period 2 of the study. The drug will be administered following a moderate calorie and fat meal. There will be a minimum washout of 7 days between each dose of study treatment.
  Interventions: Drug: GSK3640254 bis-hydrochloride salt capsule; Drug: GSK3640254 Mesylate Salt Capsule
- GSK3640254 Mesylate followed by GSK3640254 Bis-hydrochloride (Experimental): The subjects in this arm will receive an oral administration of 200 mg as 2 GSK3640254 Mesylate salt capsule (test), as single oral dose, on the morning of Day 1 during Period 1 of the study. This will be followed by an oral administration of 200 mg, as 2 GSK3640254 bis-hydrochloride salt Capsule, 100 mg (reference), as single oral dose, on the morning of Day 1 during Period 2, of the study. The drug, will be administered following a moderate calorie and fat meal. There will be a minimum washout of 7 days between each dose of study treatment.
  Interventions: Drug: GSK3640254 bis-hydrochloride salt capsule; Drug: GSK3640254 Mesylate Salt Capsule

INTERVENTIONS:
Drug: GSK3640254 bis-hydrochloride salt capsule — Administered orally (as single dose) on morning of Day 1, as 2 capsules of 100 mg following a moderate calorie and fat meal during Period 1 and Period 2, at the specified sequence, as per study.
Drug: GSK3640254 Mesylate Salt Capsule — Administered orally (as single dose) on morning of Day 1, as 2 capsules of , 100 mg following a moderate calorie and fat meal during Period 1 and Period 2, at the specified sequence, as per study.

SUMMARY:
This is a first time in human (FTIH), 2-period study, to assess the relative bioavailability of a mesylate salt capsule of GSK3640254, compared to a bis- hydrochloride salt capsule of GSK3640254, in healthy subjects, administered following a moderate calorie and fat meal. The subjects will be randomized to 2 sequences, Regimen AB or Regimen BA. For Regimen AB: The Regimen A, which will include oral administration of GSK3640254 bis-hydrochloride Capsule 200 milligram (mg) (reference), which will be administered, in Period 1 and Regimen B will include GSK3640254 Mesylate salt capsule (test), 200 mg, which will be administered in Period 2. For the regimen BA, the regimen B, will be administered, in Period 1 and regimen A, in Period 2. Each of the regimens will be given orally as 2 capsules in the morning, as per randomization sequence. There will be a minimum washout of 7 days between each dose of study treatment. A total, of 14 subjects, are planned to be enrolled in the study. The maximum duration of the study from screening to follow-up is approximately 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 to 55 years of age inclusive, at the time of signing the informed consent
* Subjects who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Body weight >= 50 kilogram (kg) for men and >= 45 kg for women, and body mass index (BMI) within the range 19.0 to 32.0 kg per meter square (kg/m^2) (inclusive).
* Male or female subjects, where a male subject must agree to use contraception, during the treatment period and for at least 14-weeks following the last dose, corresponding to the time needed to eliminate study treatment for potential genotoxic and teratogenic study treatments plus an additional 90 days (spermatogenesis cycle). In addition, male subjects must refrain from donating sperm during this period and the female subjects who is eligible to participate if she is not a woman of childbearing potential (WOCBP).
* Capable of giving signed informed consent

Exclusion Criteria:

* History of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal (GI), endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* History of clinically significant psychiatric disorders as judged by the investigator. Psychiatric disorder requiring pharmacologic treatment in the last 5 years.
* Any positive (abnormal) response confirmed by the investigator on a screening clinician (or qualified designee) administered Columbia Suicide Severity Rating Scale (CSSRS).
* History or current evidence of febrile seizures, epilepsy, convulsions, significant head injury, or other significant neurologic conditions.
* History of GI surgery (with exception of appendectomy).
* History of Cholecystectomy
* Any history of GI ulceration (esophageal, stomach, duodenal).
* Any history of GI symptoms requiring treatment in the last 3 months
* History of unexplained vaginal bleeding, endometrial hyperplasia with atypia or endometrial carcinoma
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever, is allowed unless it is active.
* ALT >1.5x upper limit of normal (ULN).
* Bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35% of total).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome).
* Medical history of cardiac arrhythmias or cardiac disease or a family or personal history of long QT syndrome.
* ECG, screening details where heart rate (<40 or >100 beats per minute [bpm]), PR interval (<120 or >220 millisecond [msec]), QRS duration (<70 or >120 msec), QT interval by Fridericia's correction formula (QTcF) interval (>450 msec) for male subjects and heart rate of <50 or >100 bpm for female subjects.
* Evidence of previous myocardial infarction (does not include ST segment changes associated with re-polarization).
* Any conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular (AV) block [2nd degree or higher], Wolf Parkinson- White [WPW] syndrome).
* Sinus Pauses >3 seconds
* Any significant arrhythmia which, in the opinion of the Investigator OR GlaxoSmithKline (GSK)/ViiV Medical monitor, will interfere with the safety for the individual subject.
* Non-sustained or sustained ventricular tachycardia (with consecutive ventricular ectopic beats).
* Prior or concomitant therapy, where past or intended use of over-the-counter or prescription medication, including herbal medications within 7 days (or 14 days if the drug is a potential enzyme inducer), or 5 half-lives (whichever is longer) prior to dosing (paracetamol/acetaminophen [up to 2 grams per day], and 2.5%, hydrocortisone [for ECG lead contact dermatitis] is permitted any time during the study).
* Prior or concurrent clinical study experience where, participation in the study would result in loss of blood or blood products in excess of 500 mL within a 56 day period; therefore donation or loss of greater than 400 mL of blood within the previous 3 months.
* Current enrollment or past participation within the last 3 months before signing of consent in this or any other clinical study involving an investigational study treatment or any other type of medical research.
* Subjects, who have previously been enrolled in this study.
* Presence of Hepatitis B surface antigen (HBsAg) at screening or positive Hepatitis C antibody test result at screening or within 3 months prior to first dose.
* Confirmed positive pre-study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV) antibody test.
* Regular use of known drugs of abuse, or history of drug or alcohol abuse in the past 5 years.
* Regular alcohol consumption within 6 months prior to the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 gram of alcohol: a half-pint (approximately 240 mL) of beer or 1 (25 mL) measure of spirits. One glass (125 mL) of wine is equivalent to 1.5 to 2 units, depending on type)
* Current use or history of regular use of tobacco- or nicotine-containing products within 6 months prior to screening. A confirmed carbon monoxide breath test reading of greater than 10 parts per million.
* Sensitivity to any of the study treatments, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening.
* Subjects who do not have the ability to swallow size 00 capsules.
* Subjects who are study site employees, or immediate family members of a study site or sponsor employee.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-08-06 (Actual); Study Completion 2018-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available, within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided, after a research proposal is submitted and has submitted approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided, for an initial period of 12 months but an extension can be granted, when justified for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Joshi SR, Fernando D, Igwe S, McKenzie L, Krishnatry AS, Halliday F, Zhan J, Greene TJ, Xu J, Ferron-Brady G, Lataillade M, Min S. Phase I evaluation of the safety, tolerability, and pharmacokinetics of GSK3640254, a next-generation HIV-1 maturation inhibitor. Pharmacol Res Perspect. 2020 Dec;8(6):e00671. doi: 10.1002/prp2.671. PMID 33200887

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single center, open-label, randomized, two-period crossover study to assess the relative bioavailability of a mesylate salt capsule of GSK3640254 compared to a hydrochloride salt capsule in healthy participants.
Pre-assignment Details: Participants received treatment in one of the two sequences; regimen A (GSK3640254 hydrochloride salt capsule) followed by regimen B (GSK3640254 mesylate salt capsule) or vice versa in each of the treatment period 1 and 2. A total of 14 participants were enrolled in the study.
Groups:
- GSK3640254 200 Mg-hydrochloride Salt Followed by Mesylate Salt: Eligible participants received a single dose of GSK3640254 200 milligram (mg) bis-hydrochloride salt (100 mg x 2 capsules) administered orally on Day 1 in treatment period 1 after a moderate fat meal. It was followed by a washout period of minimum 7 days. Participants received GSK3640254 200 mg mesylate salt (100 mg x 2 capsules) administered orally on Day 1 in treatment period 2 after a moderate fat meal.
- GSK3640254 200 Mg-mesylate Salt Followed by Hydrochloride Salt: Eligible participants received a single dose of GSK3640254 200 mg mesylate salt (100 mg x 2 capsules) administered orally on Day 1 in treatment period 1 after a moderate fat meal. It was followed by a washout period of minimum 7 days. Participants received GSK3640254 200 mg bis-hydrochloride salt (100 mg x 2 capsules) administered orally on Day 1 in treatment period 2 after a moderate fat meal.
Period: Treatment Period 1 (4 Days)
Arm/Group | GSK3640254 200 Mg-hydrochloride Salt Followed by Mesylate Salt | GSK3640254 200 Mg-mesylate Salt Followed by Hydrochloride Salt
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Washout Period (7 Days)
Arm/Group | GSK3640254 200 Mg-hydrochloride Salt Followed by Mesylate Salt | GSK3640254 200 Mg-mesylate Salt Followed by Hydrochloride Salt
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Treatment Period 2 (4 Days)
Arm/Group | GSK3640254 200 Mg-hydrochloride Salt Followed by Mesylate Salt | GSK3640254 200 Mg-mesylate Salt Followed by Hydrochloride Salt
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Eligible participants received a single dose of GSK3640254 200 mg bis-hydrochloride salt (100 mg x 2 capsules) followed by GSK3640254 200 mg mesylate salt (100 mg x 2 capsules) or vice versa, administered orally on Day 1 in each treatment period 1 and 2 following a moderate fat meal. The washout period was of minimum 7 days between the treatment periods.
Arm/Group | All Participants
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.9 (12.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 3
  White | 11

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC[0-infinity]) of GSK3640254 Following Single Oral Dose in Healthy Participants
Description: Blood samples were collected at designated timepoints. Pharmacokinetic (PK) parameters of GSK3640254 were calculated using non-compartmental methods. Geometric mean and percentage (%) geometric coefficient of variation have been presented.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48 and 72 hours post-dose in each treatment period
Population: PK Population comprising of participants in the Safety Population for whom at least one PK sample was obtained, analyzed and evaluable drug concentrations reported. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram per milliliter
Groups:
- GSK3640254 200 mg Hydrochloride Salt: Eligible participants received a single dose of GSK3640254 200 mg bis-hydrochloride salt (100 mg x 2) administered orally on Day 1 in either treatment period 1or 2 as per randomization.
- GSK3640254 Capsule 200 mg Mesylate Salt: Eligible participants received a single dose of GSK3640254 200 mg mesylate salt (100 mg x 2) administered orally on Day 1 in either treatment period 1or 2 as per randomization.
Arm/Group | GSK3640254 200 mg Hydrochloride Salt | GSK3640254 Capsule 200 mg Mesylate Salt
Number analyzed (Participants) | 14 | 14
Hour*microgram per milliliter | 23.5666 (27.2) | 27.6204 (46.7)

2. Primary Outcome: Area Under the Concentration-time Curve From Zero to Time of Last Sample Taken (AUC[0-t]) of GSK3640254 Following Single Oral Dose in Healthy Participants
Description: Blood samples were collected at designated timepoints. PK parameters of GSK3640254 were calculated using non-compartmental methods. Geometric mean and % geometric coefficient of variation have been presented. Statistical analysis of PK parameters was done using mixed effect model for evaluation of relative bioavailability (Frel). Point estimate and 90% confidence interval (CI) for the ratio of geometric least square mean of the test mesylate salt capsule to the reference Hydrochloride capsule were calculated for AUC(0-t).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, and 72 hours post-dose in each treatment period
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram per milliliter
Arm/Group | GSK3640254 200 mg Hydrochloride Salt | GSK3640254 Capsule 200 mg Mesylate Salt
Number analyzed (Participants) | 14 | 14
Hour*microgram per milliliter | 20.2797 (32.9) | 22.6494 (40.1)
Statistical Analysis 1: Comparison: GSK3640254 200 mg Hydrochloride Salt vs GSK3640254 Capsule 200 mg Mesylate Salt; Test type: Other; Ratio of geometric least square mean = 1.1169, 90% CI 2-sided [0.99 to 1.27]

3. Primary Outcome: Maximum Observed Concentration (Cmax) of GSK3640254 Following Single Oral Dose in Healthy Participants
Description: Blood samples were collected at designated timepoints. PK parameters of GSK3640254 were calculated using non-compartmental methods. Geometric mean and % geometric coefficient of variation have been presented. Statistical analysis of PK parameters was done using mixed effect model for evaluation of Frel. Point estimate and 90% CI for the ratio of geometric least square mean of the test mesylate salt capsule to the reference Hydrochloride capsule were calculated for Cmax.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, and 72 hours post-dose in each treatment period
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | GSK3640254 200 mg Hydrochloride Salt | GSK3640254 Capsule 200 mg Mesylate Salt
Number analyzed (Participants) | 14 | 14
Microgram per milliliter | 0.7357 (35.7) | 0.8502 (40.5)
Statistical Analysis 1: Comparison: GSK3640254 200 mg Hydrochloride Salt vs GSK3640254 Capsule 200 mg Mesylate Salt; Test type: Other; Ratio of geometric least square mean = 1.1556, 90% CI 2-sided [0.99 to 1.35]

4. Primary Outcome: Time to Reach Maximum Observed Concentration (Tmax) of GSK3640254 Following Single Oral Dose in Healthy Participants
Description: Blood samples were collected at designated timepoints. PK parameters of GSK3640254 were calculated using non-compartmental methods. Median and full range of Tmax have been presented.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, and 72 hours post-dose in each treatment period
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK3640254 200 mg Hydrochloride Salt | GSK3640254 Capsule 200 mg Mesylate Salt
Number analyzed (Participants) | 14 | 14
Hours | 5.0 [2 to 6] | 5.0 [2 to 6]

5. Primary Outcome: Concentration at 24 Hours Post-dose (C24h) of GSK3640254 Following Single Oral Dose in Healthy Participants
Description: Blood samples were collected at designated timepoints. PK parameters of GSK3640254 were calculated using non-compartmental methods. Geometric mean and % geometric coefficient of variation have been presented.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose in each treatment period
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | GSK3640254 200 mg Hydrochloride Salt | GSK3640254 Capsule 200 mg Mesylate Salt
Number analyzed (Participants) | 14 | 14
Microgram per milliliter | 0.3439 (37.9) | 0.3855 (45.2)

6. Secondary Outcome: Number of Participants With Non-serious Adverse Events (Non-SAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect and other situations according to medical or scientific judgement.
Time Frame: Up to 25 days
Population: Safety Population comprising of all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3640254 200 mg Hydrochloride Salt | GSK3640254 Capsule 200 mg Mesylate Salt
Number analyzed (Participants) | 14 | 14
Participants
  Any non-SAEs | 4 | 6
  Any SAEs | 0 | 0

7. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters; Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP) and Aspartate Aminotransferase (AST)
Description: Blood samples were collected to analyze the clinical chemistry parameters; ALT, ALP and AST. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the post-Dose visit value. Mean and standard deviation have been presented.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | GSK3640254 200 mg Hydrochloride Salt | GSK3640254 Capsule 200 mg Mesylate Salt
Number analyzed (Participants) | 14 | 14
International units per liter
  ALT, Day 3, n=14,14 | -1.9 (4.51) | 2.3 (6.84)
  ALP, Day 3, n=14,14 | -1.2 (7.27) | 3.0 (5.87)
  AST, Day 3, n=13,14: number analyzed (Participants) | 13 | 14
  AST, Day 3, n=13,14 | -3.5 (3.82) | -2.9 (6.55)

8. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters; Bicarbonate, Calcium, Chloride, Glucose (Fasting), Potassium, Sodium and Urea
Description: Blood samples were collected to analyze the clinical chemistry parameters; Bicarbonate, Calcium, Chloride, Glucose (fasting), Potassium, Sodium and Urea. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the post-Dose visit value. Mean and standard deviation have been presented.
Time Frame: Baseline (Day -1) and Day 3
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | GSK3640254 200 mg Hydrochloride Salt | GSK3640254 Capsule 200 mg Mesylate Salt
Number analyzed (Participants) | 14 | 14
Millimoles per liter
  Bicarbonate, Day 3, n=14,14 | -3.0 (2.66) | -2.6 (2.31)
  Calcium, Day 3, n=14,14 | -0.044 (0.1019) | 0.033 (0.0961)
  Chloride, Day 3, n=14,14 | -0.5 (1.61) | -1.7 (1.94)
  Glucose (fasting), Day 3, n=12,14: number analyzed (Participants) | 12 | 14
  Glucose (fasting), Day 3, n=12,14 | -0.17 (0.444) | 0.04 (0.554)
  Potassium, Day 3, n=14,14 | 0.21 (0.435) | 0.06 (0.445)
  Sodium, Day 3, n=14,14 | -0.9 (1.10) | -1.1 (1.56)
  Urea, Day 3, n=14,14 | -0.41 (1.634) | -0.39 (0.849)

9. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters; Bilirubin, Creatinine and Direct Bilirubin
Description: Blood samples were collected to analyze the clinical chemistry parameters; Bilirubin, Creatinine and Direct Bilirubin. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the post-Dose visit value. Mean and standard deviation have been presented.
Time Frame: Baseline (Day -1) and Day 3
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | GSK3640254 200 mg Hydrochloride Salt | GSK3640254 Capsule 200 mg Mesylate Salt
Number analyzed (Participants) | 14 | 14
Micromoles per liter
  Bilirubin, Day 3, n=14,14 | 2.1 (3.94) | -0.3 (3.81)
  Creatinine, Day 3, n=14,14 | 0.1 (7.29) | -0.1 (5.74)
  Direct Bilirubin, Day 3, n=0,1: number analyzed (Participants) | 0 | 1
  Direct Bilirubin, Day 3, n=0,1 |  | -1.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant.

10. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter; Protein
Description: Blood samples were collected to analyze the clinical chemistry parameter; Protein. Day-1 was considered as Baseline. Change from Baseline was calculated by subtracting Baseline value from the post-Dose visit value. Mean and standard deviation have been presented.
Time Frame: Baseline (Day -1) and Day 3
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | GSK3640254 200 mg Hydrochloride Salt | GSK3640254 Capsule 200 mg Mesylate Salt
Number analyzed (Participants) | 14 | 14
Grams per liter | -0.5 (3.72) | 1.4 (4.03)

11. Secondary Outcome: Number of Participants With Worst Case Hematology Results by Potential Clinical Importance (PCI) Criteria
Description: Blood samples were collected to analyze the hematology parameters; Hematocrit (Hct), Hemoglobin (Hb), Leukocytes, Lymphocytes, Neutrophils and Platelets. PCI ranges were Hct (Male and Female [high: >0.54 proportion of red blood cells in blood]), Hb (Male and Female [high: >180 grams per liter]), lymphocytes (low: <0.8x10^9 cells per liter), neutrophils (low: <1.5x10^9 cells per liter), platelets (low: <100x10^9 cells per liter and high: >550x10^9 cells per liter) and leukocytes (low: <3x10^9 cells per liter and high: >12x10^9 cells per liter). Participants were counted in the worst case category such that their value changed to (low, normal or high). If values were unchanged (example: High to High), or whose value became normal, were recorded in the 'To Normal or No Change' category.
Time Frame: Up to 22 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3640254 200 mg Hydrochloride Salt | GSK3640254 Capsule 200 mg Mesylate Salt
Number analyzed (Participants) | 14 | 14
Participants
  Hct, To low | 0 | 0
  Hct, To normal or no change | 14 | 14
  Hct, To high | 0 | 0
  Hb, To low | 0 | 0
  Hb, To normal or no change | 13 | 14
  Hb, To high | 1 | 0
  Leukocytes, To low | 0 | 0
  Leukocytes, To normal or no change | 14 | 13
  Leukocytes, To high | 0 | 1
  Lymphocytes, To low | 0 | 0
  Lymphocytes, To normal or no change | 14 | 14
  Lymphocytes, To high | 0 | 0
  Neutrophils, To low | 0 | 0
  Neutrophils, To normal or no change | 14 | 14
  Neutrophils, To high | 0 | 0
  Platelets, To low | 0 | 0
  Platelets, To normal or no change | 14 | 14
  Platelets, To high | 0 | 0

12. Secondary Outcome: Number of Participants With Urinalysis Results by Dipstick Method by Visit
Description: Urine samples were collected to assess urine bilirubin, urine glucose, urine ketones, urine leukocyte esterase (LE), urine nitrite, urine occult blood, urine protein, urobilinogen and monitor urine potential of hydrogen (pH). The dipstick test gave results in a semi-quantitative manner, and results for urinalysis parameters were recorded as negative, trace and positive, indicating proportional concentrations in the urine sample. All the numeric result values >0 have been considered as "positive".
Time Frame: Day -1 and Day 3
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3640254 200 mg Hydrochloride Salt | GSK3640254 Capsule 200 mg Mesylate Salt
Number analyzed (Participants) | 14 | 14
Participants
  Bilirubin, Day -1, Negative, n=14,14 | 14 | 14
  Bilirubin, Day -1, Trace, n=14,14 | 0 | 0
  Bilirubin, Day -1, Positive, n=14,14 | 0 | 0
  Bilirubin, Day 3, Negative, n=14,14 | 14 | 14
  Bilirubin, Day 3, Trace, n=14,14 | 0 | 0
  Bilirubin, Day 3, Positive, n=14,14 | 0 | 0
  Glucose, Day -1, Negative, n=14,14 | 14 | 14
  Glucose, Day -1, Trace, n=14,14 | 0 | 0
  Glucose, Day -1, Positive, n=14,14 | 0 | 0
  Glucose, Day 3, Negative, n=14,14 | 14 | 13
  Glucose, Day 3, Trace, n=14,14 | 0 | 0
  Glucose, Day 3, Positive, n=14,13: number analyzed (Participants) | 14 | 13
  Glucose, Day 3, Positive, n=14,13 | 0 | 0
  Ketones, Day -1, Negative, n=14,14 | 14 | 14
  Ketones, Day -1, Trace, n=14,14 | 0 | 0
  Ketones, Day -1, Positive, n=14,14 | 0 | 0
  Ketones, Day 3, Negative, n=14,14 | 14 | 14
  Ketones, Day 3, Trace, n=14,14 | 0 | 0
  Ketones, Day 3, Positive, n=14,14 | 0 | 0
  LE, Day -1, Negative, n=14,14 | 14 | 14
  LE, Day -1, Trace, n=14,14 | 0 | 0
  LE, Day -1, Positive, n=14,14 | 0 | 0
  LE, Day 3, Negative, n=14,14 | 14 | 14
  LE, Day 3, Trace, n=14,14 | 0 | 0
  LE, Day 3, Positive, n=14,14 | 0 | 0
  Nitrite, Day -1, Negative, n=14,14 | 14 | 14
  Nitrite, Day -1, Trace, n=14,14 | 0 | 0
  Nitrite, Day -1, Positive, n=14,14 | 0 | 0
  Nitrite, Day 3, Negative, n=14,14 | 14 | 14
  Nitrite, Day 3, Trace, n=14,14 | 0 | 0
  Nitrite, Day 3, Positive, n=14,14 | 0 | 0
  Occult blood, Day -1, Negative, n=14,14 | 14 | 13
  Occult blood, Day -1, Trace, n=14,14 | 0 | 0
  Occult blood, Day -1, Positive, n=14,14 | 0 | 1
  Occult blood, Day 3, Negative, n=14,14 | 14 | 14
  Occult blood, Day 3, Trace, n=14,14 | 0 | 0
  Occult blood, Day 3, Positive, n=14,14 | 0 | 0
  pH, Day -1, Negative, n=14,14 | 0 | 0
  pH, Day -1, Trace, n=14,14 | 0 | 0
  pH, Day -1, Positive, n=14,14 | 14 | 14
  pH, Day 3, Negative, n=14,14 | 0 | 0
  pH, Day 3, Trace, n=14,14 | 0 | 0
  pH, Day 3, Positive, n=14,14 | 14 | 14
  Protein, Day -1, Negative, n=14,14 | 12 | 12
  Protein, Day -1, Trace, n=14,14 | 2 | 1
  Protein, Day -1, Positive, n=14,14 | 0 | 1
  Protein, Day 3, Negative, n=14,14 | 10 | 12
  Protein, Day 3, Trace, n=14,14 | 4 | 2
  Protein, Day 3, Positive, n=14,14 | 0 | 0
  Urobilinogen, Day -1, Negative, n=14,14 | 14 | 13
  Urobilinogen, Day -1, Trace, n=14,14 | 0 | 0
  Urobilinogen, Day -1, Positive, n=14,14 | 0 | 1
  Urobilinogen, Day 3, Negative, n=14,14 | 14 | 14
  Urobilinogen, Day 3, Trace, n=14,14 | 0 | 0
  Urobilinogen, Day 3, Positive, n=14,14 | 0 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Findings for Electrocardiogram (ECG) Parameters
Description: A single 12-lead ECGs was obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, QT corrected (QTc) and QT interval corrected for heart rate according to Fridericia's formula (QTcF) intervals. Clinically significant abnormal ranges were: PR: lower: <120 milliseconds (msec) and upper: >200 msec; QRS: lower: <60 msec and upper: >120 msec and QTcF: lower: <320 msec and upper: >450 msec. The number of participants with clinically significant abnormal findings for ECG parameters have been presented.
Time Frame: Day -1, pre-dose, 2, 4, 6, 24 and 72 hours post-dose in each treatment period
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3640254 200 mg Hydrochloride Salt | GSK3640254 Capsule 200 mg Mesylate Salt
Number analyzed (Participants) | 14 | 14
Participants
  Day -1 | 0 | 0
  Pre-dose | 0 | 0
  2 hours | 0 | 0
  4 hours | 0 | 0
  6 hours | 0 | 0
  24 hours | 0 | 0
  72 hours | 0 | 0

14. Secondary Outcome: Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP) at Indicated Time-points
Description: Vital signs including DBP and SBP were measured at the indicated time-points and summarized during the study to evaluate the safety of the participants. Mean and standard deviation have been presented.
Time Frame: Day -1, pre-dose, 2, 4, 6, 24 and 72 hours post-dose in each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | GSK3640254 200 mg Hydrochloride Salt | GSK3640254 Capsule 200 mg Mesylate Salt
Number analyzed (Participants) | 14 | 14
Millimeters of mercury
  DBP, Day -1 | 64.6 (8.21) | 64.9 (8.20)
  DBP, Pre-dose | 69.4 (10.17) | 66.1 (7.64)
  DBP, 2 hours | 63.4 (7.99) | 62.7 (7.67)
  DBP, 4 hours | 65.5 (7.93) | 67.4 (8.30)
  DBP, 6 hours | 62.2 (7.83) | 63.0 (9.19)
  DBP, 24 hours | 67.2 (8.32) | 66.4 (8.63)
  DBP, 72 hours | 68.5 (6.65) | 67.7 (8.90)
  SBP, Day -1 | 118.7 (8.45) | 115.6 (9.83)
  SBP, Pre-dose | 115.9 (8.43) | 114.4 (7.97)
  SBP, 2 hours | 113.9 (8.48) | 115.1 (11.66)
  SBP, 4 hours | 112.1 (6.91) | 114.4 (9.08)
  SBP, 6 hours | 115.2 (9.93) | 116.8 (9.70)
  SBP, 24 hours | 116.1 (11.52) | 114.1 (6.89)
  SBP, 72 hours | 118.1 (8.69) | 117.4 (9.09)

15. Secondary Outcome: Pulse Rate (PR) at Indicated Time-points
Description: Vital sign including PR was measured at the indicated time-points and summarized during the study to evaluate the safety of the participants. Mean and standard deviation have been presented.
Time Frame: Day -1, pre-dose, 2, 4, 6, 24 and 72 hours post-dose in each treatment period
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK3640254 200 mg Hydrochloride Salt | GSK3640254 Capsule 200 mg Mesylate Salt
Number analyzed (Participants) | 14 | 14
Beats per minute
  Day -1 | 58.1 (7.37) | 58.4 (8.51)
  Pre-dose | 57.1 (6.90) | 56.9 (7.54)
  2 hours | 61.5 (9.45) | 60.1 (6.25)
  4 hours | 56.4 (6.69) | 57.0 (7.27)
  6 hours | 64.6 (7.08) | 66.8 (7.11)
  24 hours | 58.9 (7.90) | 58.2 (7.80)
  72 hours | 66.0 (9.47) | 64.1 (8.93)

16. Secondary Outcome: Respiratory Rate (RR) at Indicated Time-points
Description: Vital sign including RR was measured at the indicated time-point and summarized during the study to evaluate the safety of the participants. Mean and standard deviation have been presented.
Time Frame: Day -1, pre-dose, 2, 4, 6, 24 and 72 hours post-dose in each treatment period
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | GSK3640254 200 mg Hydrochloride Salt | GSK3640254 Capsule 200 mg Mesylate Salt
Number analyzed (Participants) | 14 | 14
Breaths per minute
  Day -1, n=14,14 | 15.7 (1.38) | 14.7 (1.59)
  Pre-dose, n=14,14 | 14.7 (2.20) | 15.8 (2.39)
  2 hours, n=14,14 | 15.4 (1.69) | 15.3 (0.83)
  4 hours, n=14,14 | 14.9 (1.86) | 15.2 (1.53)
  6 hours, n=14,14 | 14.8 (1.37) | 15.8 (1.12)
  24 hours, n=13,14: number analyzed (Participants) | 13 | 14
  24 hours, n=13,14 | 14.2 (2.08) | 15.4 (1.16)
  72 hours, n=14,14 | 14.8 (1.97) | 13.9 (2.57)

17. Secondary Outcome: Temperature at Indicated Time-points
Description: Vital sign including temperature was measured at the indicated time-points and summarized during the study to evaluate the safety of the participants. Mean and standard deviation have been presented.
Time Frame: Day -1, pre-dose, 2, 4, 6, 24 and 72 hours post-dose in each treatment period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | GSK3640254 200 mg Hydrochloride Salt | GSK3640254 Capsule 200 mg Mesylate Salt
Number analyzed (Participants) | 14 | 14
Celsius
  Day -1 | 36.74 (0.227) | 36.67 (0.133)
  Pre-dose | 36.63 (0.120) | 36.59 (0.103)
  2 hours | 36.66 (0.115) | 36.64 (0.115)
  4 hours | 36.66 (0.109) | 36.63 (0.144)
  6 hours | 36.64 (0.140) | 36.69 (0.141)
  24 hours | 36.67 (0.120) | 36.64 (0.074)
  72 hours | 36.74 (0.165) | 36.79 (0.228)

18. Secondary Outcome: Number of Participants With the Indicated Assessment Events of Suicidal Behavior (SB) and Suicidal Ideation (SI) Via the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: Assessment of suicidality was conducted using the C-SSRS, a brief questionaire designed to assess severity and change in suicidality by integrating both behavior and ideation using a semi-structured interview to probe participant responses.
Time Frame: Day 3 in each treatment period
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3640254 200 mg Hydrochloride Salt | GSK3640254 Capsule 200 mg Mesylate Salt
Number analyzed (Participants) | 14 | 14
Participants
  SI- Wish to be dead | 0 | 0
  SI- Non-specific (no method, intent or plan) | 0 | 0
  SI- Method, but no intent or plan | 0 | 0
  SI- Method and intent, but no plan | 0 | 0
  SI- Method, intent, and plan | 0 | 0
  SB- Preparatory acts or behaviour | 0 | 0
  SB- Aborted attempt | 0 | 0
  SB- Interrupted attempt | 0 | 0
  SB- Non-fatal actual suicide attempt | 0 | 0
  SB- Completed suicide | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs and non-serious AEs were collected from the start of study treatment up to 25 days.
Description: SAEs and Non-SAEs were reported by treatment for the Safety Population which comprised of all randomized participants who received at least 1 dose of study treatment.
Arm/Group | GSK3640254 200 mg Hydrochloride Salt | GSK3640254 Capsule 200 mg Mesylate Salt
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 3/14 | 6/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3640254 200 mg Hydrochloride Salt (N=14) | GSK3640254 Capsule 200 mg Mesylate Salt (N=14)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-05-29): https://cdn.clinicaltrials.gov/large-docs/62/NCT03575962/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT03575962/SAP_001.pdf